CLINICAL TRIAL: NCT04123626
Title: A Prospective First-In-Human Study to Evaluate the Safety and Tolerability of QR-1123 in Subjects With Autosomal Dominant Retinitis Pigmentosa (adRP) Due to the P23H Mutation in the RHO Gene
Brief Title: A Study to Evaluate the Safety and Tolerability of QR-1123 in Subjects With Autosomal Dominant Retinitis Pigmentosa Due to the P23H Mutation in the RHO Gene
Acronym: AURORA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ProQR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PQ-1123-001
Record Dates: First submitted 2019-10-01; First posted 2019-10-11 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Autosomal Dominant Retinitis Pigmentosa; Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Disease; Retinitis; Vision Tunnel; Vision Disorders
Keywords: adRP; Retinitis Pigmentosa; P23H mutation; Rhodopsin; antisense oligonucleotide; IVT; autosomal dominant
MeSH Terms: conditions — Eye Diseases; Eye Diseases, Hereditary; Retinal Dystrophies; Retinal Diseases; Retinitis; Vision Disorders; Retinitis Pigmentosa; Night Blindness, Congenital Stationary, Autosomal Dominant 1; Multiple Pterygium Syndrome, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single dose cohorts are open label. Repeat dose cohorts are randomized, double masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- QR-1123 Single dose - dose level 1 (Experimental): Open label Single dose cohort: dose level 1
  Interventions: Drug: QR-1123
- QR-1123 Single dose - dose level 2 (Experimental): Open label Single dose cohort: dose level
  Interventions: Drug: QR-1123
- QR-1123 Single dose - dose level 3 (Experimental): Open label Single dose cohort: dose level 3
  Interventions: Drug: QR-1123
- QR-1123 Single dose - dose level 4 (Experimental): Open label Single dose cohort: dose level 4
  Interventions: Drug: QR-1123
- QR-1123 Single dose - dose level 5 (Experimental): Open label Single dose cohort: dose level 5
  Interventions: Drug: QR-1123
- Repeat dose cohort 1 (Experimental): Double-masked, randomized, sham controlled, Repeat dose cohort. Dose levels will be determined following DMC review of obtained safety and efficacy data.
  Interventions: Drug: QR-1123; Other: Sham procedure

INTERVENTIONS:
Drug: QR-1123 — unilateral IVT injection
Other: Sham procedure — Sham procedures (i.e. no penetration of the globe) closely mimic the active injection and serve to mask subjects to treatment assignment
  Arms: Repeat dose cohort 1

SUMMARY:
This study evaluates the safety, tolerability and efficacy of QR-1123 injection in the eye (intravitreal; IVT) injections (one eye/unilateral) in subjects receiving a single dose or repeat doses. Single injections will be assessed in an open label way, and repeat injections will be assessed in a double-masked, randomized, sham-controlled fashion.

DETAILED DESCRIPTION:
QR-1123 is an antisense oligonucleotide, designed to specifically target the mutant P23H messenger ribonucleic acid (mRNA) in order to reduce the expression of the P23H protein selectively, while preserving expression of the wild type (WT) rhodopsin (RHO) protein. It is hypothesized that the reduction of mutant P23H mRNA will reduce the deleterious effects of the dominant-negative protein and should result in increased function of WT rhodopsin protein in photoreceptors. Restoration of WT RHO function is expected to improve vision in patients with adRP due to the P23H mutation.

The study will comprise up to 8 single dose and repeat dose cohorts. Prior to initiating a higher single dose cohort and/or prior to initiating repeat dose cohort(s), available safety and efficacy data will be reviewed by the DMC.

In the single dose cohorts subjects will receive a single, unilateral IVT injection of QR-1123 in an open label fashion. In the repeat dose cohorts subjects will be randomized to receive either a unilateral IVT injection of QR-1123 every 3 months or a unilateral sham procedure every 3 months, in a double masked fashion. Subjects will be followed for safety, tolerability and efficacy for a total period of 12 months.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female, ≥ 18 years of age.
2. Clinical presentation consistent with adRP, based on ophthalmic examinations.
3. Impairment on VF in the opinion of the Investigator, as determined by perimetry.
4. A molecular diagnosis of autosomal dominant form of RP with the P23H mutation in the RHO gene, based on genetic analysis.
5. A clear ocular media and adequate pupillary dilation to permit good quality fundus imaging, as assessed by the Investigator.

Main Exclusion Criteria:

1. Presence of additional pathogenic mutations in genes (other than the P23H mutation in the RHO gene) associated with inherited retinal degenerative diseases or syndromes, based on genetic analysis (eg, Usher syndrome, Leber congenital amaurosis, etc).
2. Presence of any significant ocular or non-ocular disease/disorder (including medication and laboratory test abnormalities) which, in the opinion of the Investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or the subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-06-07 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of ocular AEs | up to 12 months
  Incidence and severity of ocular adverse events scored based on CTCAC in the study and fellow eye
Incidence and Severity of non-ocular AEs | up to 12 months
  Incidence and severity of non-ocular adverse events scored based on CTCAC in the study and fellow eye

SECONDARY OUTCOMES:
Changes in BCVA | up to 12 months
  Changes in Best corrected visual acuity (BCVA)
Changes in LLVA | up to 12 months
  Changes in Low-luminance visual acuity (LLVA)
Changes in DAC perimetry | up to 12 months
  Changes in Dark adapted chromatic (DAC) perimetry
Changes in Static VF | up to 12 months
  Changes in Static VF (Visual Field)
Changes in Microperimetry | up to 12 months
  Changes in Microperimetry
Changes in SD-OCT | up to 12 months
  Changes in Spectral Domain-Optical Coherence Tomography
Changes in FST | up to 12 months
  Changes in Full-field Stimulus Threshold (FST)
Changes in Full-field ERG | up to 12 months
  Changes in Full-field Electroretinogram (ERG)
Assessment of systemic exposure after treatment with QR-1123 | up to 12 months
  Serum levels of QR-1123

CONTACTS AND LOCATIONS:
Overall Officials: ProQR Medical Monitor, Study Director — ProQR Therapeutics; ProQR Clinical Trial Manager, Study Director — ProQR Therapeutics
Locations (5):
- United States (5):
  - Sue Anschutz-Rogers Eye Center, University of Colorado - Dept. of Ophthalmology, Aurora, Colorado
  - VitreoRetinal Associates, Gainesville, Florida
  - Shriners UK Ophthalmology - University of Kentucky, Lexington, Kentucky
  - Casey Eye Institute, OHSU, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided